CLINICAL TRIAL: NCT03579732
Title: EffectiveNess of Low Dose Aspirin in GastrointEstinal Cancer Prevention - Taiwan
Acronym: ENgAGE-Taiwan
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 19882
Record Dates: First submitted 2018-06-26; First posted 2018-07-09 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Colorectal Neoplasms
Keywords: Low-dose aspirin,; Cancer prevention
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Aspirin; N-acetyl-S-(alpha-methyl-4-(2-methylpropyl)benzeneacetyl)cysteine 4-(nitrooxy)butyl ester

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Long-term users: Adults using low-dose aspirin for > 3 years
  Interventions: Drug: Aspirin (Acetylsalicylic Acid, BAYE4465)
- Episodic users: Adults using low-dose aspirin inconsistently, or consistently but < 3 years
  Interventions: Drug: Aspirin (Acetylsalicylic Acid, BAYE4465)
- Former users: Subset of adult Episodic users of aspirin who discontinued the drug for at least 1 year before case/ control date
  Interventions: Drug: Aspirin (Acetylsalicylic Acid, BAYE4465)
- Non-consumers: Adults who did not use low-dose aspirin
  Interventions: Other: No drug

INTERVENTIONS:
Drug: Aspirin (Acetylsalicylic Acid, BAYE4465) — Low dose of aspirin, i.e. < 150 mg daily
  Groups: Episodic users; Former users; Long-term users
Other: No drug — Non-consumers
  Other Names: No aspirin
  Groups: Non-consumers

SUMMARY:
The study evaluates the protective effect of low-dose aspirin use on gastrointestinal cancers (colorectal, esophageal and gastric cancers) in long-term users, episodic users and non-users of aspirin in Taiwan.

DETAILED DESCRIPTION:
The primary objective is to investigate the protective effect of long-term low dose use of aspirin on colorectal, esophageal and gastric cancer in adult subjects from Taiwan.

Secondary objectives are to evaluate the protective effect by duration of low-dose aspirin use on colorectal cancer, the effect of discontinuation of aspirin on colorectal cancer prevention, the staging distribution of colorectal cancer and the description of fatal cases due to colorectal cancer.

Aspirin use will be identified through Taiwanese National Health Insurance (NIH) data from 2000 to 2015. Cancer cases and staging of the three cancer types will be ascertained through the Taiwan Cancer Registry, using data from 2000 to 2014. Fatal cases will be ascertained using Mortality database from 2000 to 2015.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 or older at the cohort entry date.
* Taiwanese National Health Insurance enrollees with non-missing and consistent age and gender information.

Exclusion Criteria:

* Subjects with any cancer diagnosis before cohort entry date.
* No use of National Health Insurance before the cohort entry date.
* Low dose aspirin prescription before cohort entry date.
* Subjects with conditions contra-indicated for low dose aspirin use before cohort entry date.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be selected from the Taiwanese National Health Insurance (NIH) database.
Sampling Method: Non-Probability Sample
Enrollment: 4710504 (Actual)
Dates: Start 2018-06-29 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Number of subjects with colorectal cancer | Up to 14 years
  Number of subjects with colorectal cancer for each cohort (long-term, episodic and former users of aspirin, and non-users).
Number of subjects with esophageal cancer | Up to 14 years
  Number of subjects with esophageal cancer for each cohort (long-term, episodic and former users of aspirin, and non-users).
Number of subjects with gastric cancer | Up to 14 years
  Number of subjects with gastric cancer for each cohort (long-term, episodic and former users of aspirin, and non-users).

SECONDARY OUTCOMES:
Duration of aspirin use to colorectal cancer | Up to 14 years
  The duration of low-dose aspirin use in years to colorectal cancer.
Time from aspirin discontinuation to colorectal cancer | Up to 14 years
  Period of time in years from discontinuation of aspirin use to detection of colorectal cancer.
Stage of colorectal cancer | Up to 14 years
  The stage of cancer will be determined according to the International Classification of Diseases for Oncology (ICD-O-3).
Number of fatal cases due to colorectal cancer | Up to 14 years
  Derived from Taiwan Mortality database.

CONTACTS AND LOCATIONS:
Locations (1):
- National University of Taiwan Hospital, Taipei, Taiwan